CLINICAL TRIAL: NCT01220050
Title: A PROSPECTIVE, PILOT, CROSS-OVER STUDY TO ASSESS THE EFFICACY OF PARICALCITOL IN REDUCING PARATHYROID HORMONE LEVELS AND AMELIORATING MARKERS OF BONE REMODELLING IN RENAL TRANSPLANT RECIPIENTS WITH SECONDARY HYPERPARATHYROIDISM
Brief Title: Paricalcitol in Reducing Parathyroid Hormone Levels and Ameliorating Markers of Bone Remodelling in Renal Transplant Recipients With Secondary Hyperparathyroidism
Acronym: APPLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APPLE; 2008-006380-36 (EudraCT Number)
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Renal Transplant; Secondary Hyperparathyroidism
Keywords: Paricalcitol; Renal transplant; Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — paricalcitol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol (Experimental)
  Interventions: Drug: Paricalcitol
- Standard therapy (Active Comparator)
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol capsules 1- 2 mcg/day/pts for 26 weeks
  Arms: Paricalcitol
Drug: Standard therapy — Standard therapy for hyperparathyroidism for 26 weeks
  Arms: Standard therapy

SUMMARY:
The risk of fracture for kidney transplant recipients is 4 times higher that of the general population. The hyperparathyroidism plays a key role in the maintenance or development of post-transplant alterations of bone remodelling.

Renal transplant patients are at high risk of hyperparathyroidism, largely because of long-lasting renal insufficiency before transplant, and of progressive deterioration of kidney function because of chronic allograft nephropathy (a disease of proteinuria and progressive decline of the glomerular filtration rate).In hemodialysis patients, intravenous paricalcitol (19-nor-1,25-dihydroxyvitamin D2), a new vitamin D analogue, achieves a faster and more effective normalization of parathyroid hormone (PTH) levels than calcitriol (1,25-dihydroxyvitamin D3), an effect that is associated with smaller changes in serum calcium and phosphorus levels.

Whether oral paricalcitol may help achieving a prompt reduction in serum PTH levels and, secondarily, in urinary protein excretion in renal transplant recipients with secondary hyperparathyroidism is worth investigating.

DETAILED DESCRIPTION:
BACKGROUND The risk of fracture for kidney transplant recipients is 4 times higher that of the general population. The pathogenesis of post-transplant bone disease is multifactorial, but hyperparathyroidism plays a key role in the maintenance or development of post-transplant alterations of bone remodelling. Vitamin D and its analogues are key components of treatment aimed to prevent or ameliorate secondary hyperparathyroidism in patients with chronic kidney disease (CKD). In hemodialysis patients, intravenous paricalcitol (19-nor-1,25-dihydroxyvitamin D2), a new vitamin D analogue, achieves a faster and more effective normalization of parathyroid hormone (PTH) levels than calcitriol (1,25-dihydroxyvitamin D3), an effect that is associated with smaller changes in serum calcium and phosphorus levels. Preliminary evidence is also available that in pre-dialysis patients with CKD and secondary hyperparathyroidism, treatment with oral paricalcitol may also reduce urinary protein excretion, an effect that is independent of concomitant treatment with agents that block the renin-angiotensin system and that in the long-term might translate into slower progression to end stage kidney disease and need for renal replacement therapy.

Renal transplant patients are at high risk of hyperparathyroidism, largely because of long-lasting renal insufficiency before transplant, and of progressive deterioration of kidney function because of chronic allograft nephropathy (a disease of proteinuria and progressive decline of the glomerular filtration rate). Whether oral paricalcitol may help achieving a prompt reduction in serum PTH levels and, secondarily, in urinary protein excretion in renal transplant recipients with secondary hyperparathyroidism is worth investigating.

AIMS Primary To evaluate whether 6-months treatment with paricalcitol may achieve a prompt and effective reduction in PTH serum levels in stable renal transplant patients with secondary hyperparathyroidism.

DESIGN This will be a Prospective, Randomized, Open label, Cross-over study of 6-months with Paricalcitol or standard treatment for hyperparathyroidism.

After one month wash-out from any form of Vitamin D therapy, patients satisfying the inclusion/exclusion criteria will be randomized to two treatment arms:

1. Paricalcitol capsules 1- 2 mcg/day/pts for 26 weeks
2. Standard therapy for hyperparathyroidism for 26 weeks At the end of the first treatment period with Paricalcitol or Standard therapy each patient will cross-over to the other treatment.

After baseline evaluation eligible patients will enter a 6 months treatment period whit oral paricalcitol (1-2 mcg/day), or standard treatment for hyperparathyroidism, added-on background therapy whit calcium and phosphate supplementation as deemed clinically appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >18 years old
* Renal transplant recipients with persistent secondary hyperparathyroidism
* PTH persistently >80 pg/mL up 2 month post transplant (stable or progressively increasing PTH levels)
* No ongoing therapy with Vitamin D
* Patients on maintenance therapy with calcineurin inhibitors and Mycophenolate Mofetil or Azathioprine
* Serum creatinine < 2mg/dL
* Patients legally able to give written informed consent to the trial (signed and dated by the patient)
* Written informed consent.

Exclusion Criteria:

* Concomitant administration of other forms of Vitamin D (different from paricalcitol)
* PTH< 80 pg/ml
* Serum Ca> 10,2 mg/dL
* Clinically serious condition
* History of malignancy
* Evidence of active hepatitis C virus, hepatitis B virus or human acquired immunodeficiency virus infection
* Specific contraindications or history of hypersensitivity to the study drugs;
* Previous history of allergy or intolerance, or evidence of immunologically-mediated renal disease, systemic diseases, cancer
* Drug or alcohol abuse
* Any chronic clinical conditions that may affect completion of the trial or confound data interpretation
* Pregnancy or lactating
* Women of childbearing potential without following a scientifically accepted form of contraception
* Legal incapacity
* Evidence of an uncooperative attitude
* Any evidence that patient will not be able to complete the trial follow-up.
* Previous diagnosis of: intellectual disability/mental retardation, dementia, schizophrenia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
PTH reduction during the 6 months of paricalcitol therapy (during both treatment periods) compared to the change in PTH levels during the corresponding 6 months without paricalcitol therapy. | Every three months.

SECONDARY OUTCOMES:
Measurement of osteocalcin. | Baseline and then every three months.
Measurement of bone alkaline phosphatase. | Baseline and then every three months.
Measurement of urinary deoxypyridinoline. | Baseline and then every three months.
Bone mineral density (by MOC). | At baseline and at the end of both treatment periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Negri Institute - Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy